CLINICAL TRIAL: NCT03864900
Title: Efficacy of a Health Belief Model Based Intervention for Anticoagulation Adherence in Patients With Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: Efficacy of a Health Belief Model Based Intervention for Anticoagulation Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Taipei Medical University WanFang Hospital (Other); Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, RN PhD Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 201505054
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Anticoagulants
Keywords: Anticoagulants; Atrial fibrillation; Adherence; Health belief model
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The health belief model based medication adherence intervention comprised two main components: a 60-minute individual face to face instruction and six follow-up telephone calls.
Who Masked: Participant, Care Provider
Masking Description: Both participants and care providers were unaware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The medication adherence intervention comprised two main components: a 60-minute individual face to face instruction and six follow-up telephone calls.
  Interventions: Behavioral: The medication adherence intervention
- The control group (No Intervention): Participants in the control group received regular medication education, 10-minute individual instruction for health knowledge and six follow-up telephone calls for concerning health.

INTERVENTIONS:
Behavioral: The medication adherence intervention — The health belief model based medication adherence intervention comprised two main components: a 60-minute individual face to face instruction and six follow-up telephone calls.
  Arms: The intervention group

SUMMARY:
Inconsistent anticoagulation therapy in AF patients is associated with a higher risk of stroke and abnormal bleeding. The purpose of the study is to investigate the efficacy of a health belief model based self-management of oral anticoagulant therapy intervention on the outcome of medication adherence and the mediators of knowledge, professional support, health belief, and self-efficacy in patients treated with oral anticoagulants for atrial fibrillation. A randomized clinical trial with repeated measurements was conducted. A convenient sample of 110 adults who were treated with anticoagulants for atrial fibrillation was recruited from two teaching hospitals in northern Taiwan. Participants were randomly assigned 1:1 to either the control group (n = 36) or the intervention group (n = 36) after completion of baseline questionnaires. Patients in the experimental group received the health belief model based anticoagulation adherence intervention, including one 60-minute individual instructions and six 15-minute telephone follow-ups. Participants in the control group received regular medication education, 10-minute individual instruction for health knowledge and six follow-up telephone calls for concerning health. Patients in both groups answered the study questionnaires at three and six months. The generalized estimating equations were used to analyze the efficacy of the intervention for enhancing knowledge, knowledge, perceived benefits, perceived barriers, self-efficacy, and adherence to anticoagulant therapies in patients treated with oral anticoagulants for atrial fibrillation. The results of the study will contribute to the knowledge for improving adherence to oral anticoagulation therapies in patients with atrial fibrillation.

DETAILED DESCRIPTION:
BACKGROUND: Inconsistent anticoagulation therapy in AF patients is associated with a higher risk of stroke and abnormal bleeding. However, control of oral anticoagulation therapy in AF patients has been frequently reported as inadequate. Few theoretical based interventions have been tested for enhancing medication adherence in this population. Previous studies showed that the health belief model may offer some advantage over other behavior change theories for enhancing medication adherence in adult with chronic conditions.

PURPOSE: The purpose of the study is to investigate the efficacy of a health belief model based self-management of oral anticoagulant therapy intervention on the outcome of medication adherence and the mediators of knowledge, professional support, health belief, and self-efficacy in patients treated with oral anticoagulants for atrial fibrillation.

METHODS: The study is a randomized clinical trial with repeated measurements. A convenient sample of 72 adults who were treated with anticoagulants for atrial fibrillation was recruited from two teaching hospitals in northern Taiwan. Participants were randomly assigned 1:1 to either the control group (n = 36) or the intervention group (n = 36) after completion of baseline questionnaires. Allocation was balanced by site by using a minimization method. The health belief model based self-management intervention comprised two main components: a 60-minute individual face to face instruction and six follow-up telephone calls. Participants in the control group received regular medication education, 10-minute individual instruction for health knowledge and six follow-up telephone calls for concerning health. Data were collected at baseline, third month, and sixth month in both groups, by using self-administered questionnaires. The investigator administered the study questionnaire after obtaining informed consent from each subject. The data collection took place at the waiting areas outside the outpatient clinics during the patients' visits to the clinics. For subjects who were unable to read the questionnaire due to vision or other problems, the investigator read each question to help them complete the questionnaire. The instruments include the Atrial Fibrillation Knowledge Scale, Satisfaction Scale about Service and Warfarin Treatment, Belief About Anticoagulation Survey, and Self-Efficacy for Appropriate Medication Use Scale.

DATA ANALYSIS: Data were analyzed using the Statistical Package for Social Sciences 20.0 (SPSS, Inc., Chicago, IL, USA). Descriptive analyses were used to describe study variables. Independent t-tests and one-way analysis of variance (ANOVA) were performed to analyze the baseline equivalent between study groups. The generalized estimating equations were used to analyze the efficacy of the intervention for enhancing knowledge, knowledge, perceived benefits, perceived barriers, self-efficacy, and adherence to anticoagulant therapies in patients treated with oral anticoagulants for atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20 years of age
2. fluent in Mandarin or Taiwanese
3. diagnosed with AF
4. treated with warfarin or NOACs for anticoagulation.

Exclusion Criteria:

1. diagnosed with psychological diseases
2. diagnosed with uncontrolled hypertension
3. diagnosed with the New York Heart Association (NYHA) grade VI heart failure
4. implanted with a cardiac pacemaker
5. had cardiac surgery in the past three months
6. hospitalized for AF in the past three months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsae Jyy Wang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (2):
- Taiwan (2):
  - Taipei Medical University Shuang Ho Hospital, Taipei County, Taipei
  - Taipei Medical University WanFang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiang CE, Wu TJ, Ueng KC, Chao TF, Chang KC, Wang CC, Lin YJ, Yin WH, Kuo JY, Lin WS, Tsai CT, Liu YB, Lee KT, Lin LJ, Lin LY, Wang KL, Chen YJ, Chen MC, Cheng CC, Wen MS, Chen WJ, Chen JH, Lai WT, Chiou CW, Lin JL, Yeh SJ, Chen SA. 2016 Guidelines of the Taiwan Heart Rhythm Society and the Taiwan Society of Cardiology for the management of atrial fibrillation. J Formos Med Assoc. 2016 Nov;115(11):893-952. doi: 10.1016/j.jfma.2016.10.005. Epub 2016 Nov 24. PMID 27890386
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Alexandru Popescu B, Schotten U, Van Putte B, Vardas P. 2016 ESC Guidelines for the Management of Atrial Fibrillation Developed in Collaboration With EACTS. Rev Esp Cardiol (Engl Ed). 2017 Jan;70(1):50. doi: 10.1016/j.rec.2016.11.033. No abstract available. English, Spanish. PMID 28038729
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The Intervention Group | The Control Group
Started | 36 | 36
Completed | 33 | 30
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — medical reason: change anticoagulation drug, Hemorrhage, operation | 2 | 5

BASELINE CHARACTERISTICS:
Population: Age 20 years and over, diagnosed with AFib by physical and receiving anticoagulation therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | The Intervention Group | The Control Group | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (7.5) | 73.3 (10) | 71.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 24 | 19 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 36 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 36 | 36 | 72
Kinds of Anticoagulation [Number; unit: participants]
  Warfarin | 17 | 17 | 34
  NOACs | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: The Short-form Adherence to Reﬁlls and Medications Scale (ARMS)
Description: There are seven items in the scale. Subjects were asked to indicate how often they actually miss taking their anticoagulants in each item on a 4-point Likert scale (1_ none of the time to 4_ all of the time). The total score of the 7 items represents the scale score, with a possible range of 7 to 28. A higher score indicates worse adherence to anticoagulation treatment.
Time Frame: baseline (T1), 12th week (T2), and 24th week (T3) follow-ups.
Population: All participants with baseline and at least fellow up for 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Intervention Group | The Control Group
Number analyzed (Participants) | 36 | 36
score on a scale
  baseline (T1) | 9.6 (1.6) | 9.4 (1.7)
  12th week (T2) | 8.5 (1.7) | 9.3 (2.2)
  24th week (T3) | 8.1 (1.4) | 9.2 (2.2)

2. Secondary Outcome: The Knowledge of Warfarin Anticoagulation Treatment Scale
Description: The 11-item scale covers four areas of warfarin treatment knowledge: administration (e.g., dose, color, and route of administration), interaction with foods, interaction with other drugs, and side effects. There are five choices for each item, and only one of the choices is correct (scored 1). The total score of the 11 items represents the scale score, with a possible range of 0 to 11. Higher scores indicate higher levels of understanding of warfarin treatment. The scale was also modified to measure the NOACs treatment knowledge. To facilitate analysis and comparison, the score of each scale was converted to a scale of 0 to 100 (actual score/possible maximum score x 100).
Time Frame: baseline (T1), 12th week (T2), and 24th week (T3) follow-ups.
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Arm/Group | The Intervention Group | The Control Group
Number analyzed (Participants) | 36 | 36
percentage of accuracy
  Baseline (T1) | 35.9 (15.7) | 36.9 (20.0)
  12th week (T2) | 63.9 (22.5) | 43.7 (23.0)
  24th week (T3) | 66.4 (18.2) | 49.5 (21.8)

3. Secondary Outcome: The Perceived Benefits Subscale of the Beliefs About Anticoagulation Survey (BAAS)
Description: The subscale covers 5 potential benefits of taking anticoagulation, including lessening the risk of having a stroke, lowering the chance of being hospitalized, feeling healthier, improving quality of life, and worrying less about the disease. For each item, the subjects indicated their levels of agreement on a 5-point Likert scale (from 1_ strongly disagree to 5_ strongly agree). The potential scores range from 5 to 25 points, with higher scores indicating higher levels of perceived benefits associated with taking anticoagulation.
Time Frame: baseline (T1), 12th week (T2), and 24th week (T3) follow-ups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The Intervention Group | The Control Group
Number analyzed (Participants) | 36 | 32
units on a scale
  baseline (T1) | 20.2 (2.6) | 19.9 (2.0)
  12th week (T2) | 20.9 (2.6) | 19.8 (1.3)
  24th week (T3) | 21.6 (2.6) | 20.3 (2.1)

4. Secondary Outcome: The Concerns About Anticoagulation Therapy Scale
Description: The scale lists ten potential concerns, including drug interactions, forgetting to take anticoagulants, side effects, hospital visits, diet interactions, activity restrictions, impact on work, not helpful, and difficulty of following instructions. The subjects were asked to indicate all concerns that apply to them. Each concern was scored 1. The potential scores range from 0 to 10, with higher scores indicating more concerns.
Time Frame: baseline (T1), 12th week (T2), and 24th week (T3) follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Intervention Group | The Control Group
Number analyzed (Participants) | 36 | 36
score on a scale
  baseline (T1) | 1.2 (1.4) | 1.8 (1.4)
  12th week (T2) | 0.8 (1.4) | 1.4 (1.5)
  24th week (T3) | 0.5 (1.0) | 1.1 (1.2)

5. Secondary Outcome: The Self-efficacy for Appropriate Medication Use Scale (SEAMS)
Description: The 13-item scale covers two dimensions of self-efficacy: for taking medications under difficult circumstances and for taking medications under uncertain or changing circumstances. For each item, the subjects indicated their level of confidence about taking medications correctly under a specific circumstance on a three-point response scale (1 _ not confident, 2 _ somewhat confident, and 3 _ very confident). The potential scores range from 13 to 39, with high scores indicating higher levels of self-efficacy for appropriate anticoagulant use.
Time Frame: baseline (T1), 12th week (T2), and 24th week (T3) follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Intervention Group | The Control Group
Number analyzed (Participants) | 36 | 36
score on a scale
  baseline (T1) | 32.0 (6.0) | 31.4 (6.4)
  12th week (T2) | 33.7 (5.2) | 33.1 (5.5)
  24th week (T3) | 35.3 (4.5) | 33.3 (4.6)

6. Other Pre Specified Outcome: The Satisfaction Scale About Service and Warfarin Treatment (SSWT)
Description: The original scale includes seven positive statements about the services and warfarin treatment. In the current study, the term of warfarin was replaced with anticoagulants. The item 5 (regarding INR monitoring) in the original scale was deleted as it only applies to patients treated with warfarin. Therefore, there were only six items used in the current study. For each item, the subjects indicated their levels of agreement on a 5-point Likert scale (from 0_ strongly disagree to 4_ strongly agree). The total score of the 6 items represents the scale score, with a possible range of 0 to 24. Higher scores indicate higher levels of satisfaction about service and warfarin treatment.
Time Frame: baseline (T1), 12th week (T2), and 24th week (T3) follow-ups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Intervention Group | The Control Group
Number analyzed (Participants) | 36 | 36
score on a scale
  baseline (T1) | 19.7 (3.1) | 18.8 (2.9)
  12th week (T2) | 19.4 (2.9) | 18.9 (2.6)
  24th week (T3) | 20.6 (3.0) | 19.7 (3.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | The Intervention Group | The Control Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT03864900/Prot_SAP_000.pdf